CLINICAL TRIAL: NCT04733716
Title: Tourniquet Use Does Not Affect Pain and Function After Total Knee Arthroplasty: Patient Evaluation According to Pain Threshold
Brief Title: Does Tourniquet Use Have an Effect on Pain and Function After Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Savaş Çamur, Principal Investigator, Umraniye Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2020/13
Record Dates: First submitted 2021-01-26; First posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Arthropathy of Knee; Pain, Joint
Keywords: Knee Arthroplasty
MeSH Terms: conditions — Arthralgia

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The pain sensitivity of all measurement patients was taken on the day before the surgery by the same author, and these values were blinded from another author who recorded the repetitive postoperative VAS and knee scores.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total Knee Arthroplasty with using Tourniquet (Active Comparator): A pneumatic tourniquet was used before surgery at the proximal thigh and inflated before the skin incision until skin closure in this group. The tourniquet was inflated to either 275 or 325 mmHg, depending on the patient's systolic blood pressure.
  Interventions: Procedure: Using Tourniquet
- Total Knee Arthroplasty without using Tourniquet (Active Comparator): A pneumatic tourniquet was not used in this group during the total knee arthroplasty.
  Interventions: Procedure: Using Tourniquet

INTERVENTIONS:
Procedure: Using Tourniquet — The purpose of this prospective randomized double blinded study was to compare the effect of using a tourniquet on early-stage pain and 1-year postoperative functional outcomes when patients were divided into two groups according to the pain threshold.

SUMMARY:
Total knee arthroplasty (TKA) is an effective surgical procedure for reducing knee joint pain and improving the quality of life of patients with advanced knee osteoarthritis. Although advanced surgical techniques and prosthesis design are achieved, postoperative pain is a significant factor that affects those patients who have undergone TKA with a satisfactory outcome. The reasons for postoperative pain after TKA are somewhat unclear Although there are studies evaluating the preoperative and postoperative conditions of the patients using pain scores, these values differ greatly in patients who are suitable for the same procedure. Previous studies have demonstrated that variability exists between individuals in basal pain sensitivity, which is assessed using quantitative sensory testing To our knowledge, only one study has investigated the pain condition using an algometer and postoperative pain and the analgesic requirement on the day of surgery and during the postoperative period.Unlike the above-cited study, in this study, we evaluated the effect of using a tourniquet on early-stage pain and 1-year postoperative functional outcomes when patients were divided into two groups according to the pain threshold.

DETAILED DESCRIPTION:
This is a prospective double-blinded, randomized controlled trial diagnostic study conducted at a single center from June 2018 to December 2019. Patients who underwent total knee arthroplasty due to end-stage knee osteoarthritis were asked to volunteer to participate in this study. A prospective randomized study was conducted using a digital algometer to assess the pain sensitivity for the relationship between postoperative early-stage pain score and first-year functional scores in patients with or without using tourniquet who underwent primary TKA. Patients were randomized to with or without tourniquet groups; a random number generated by the research staff determined the group designation, independent of a senior surgeon. T All participants in this study gave their written informed consent. Patients with a neurological disorder, diagnosed with fibromyalgia, history of knee operation, valgus knee, greater than 30° flexion contracture that had undergone bilateral knee arthroplasty or revision knee arthroplasty, chronic analgesic users, and those with a psychiatric disease were excluded from this study.

Preoperative Procedure: All patients had anterior-posterior and lateral radiographs of the bilateral knees, taken with a standard full-length weight-bearing the patients in bipedal stance, the knees in maximal extension for anterior-posterior and 30-degree flexion for lateral radiographs pre and postoperatively. In all patients, range of motion and contractures of both knee joints were recorded. All patient's educational level was also assessed. The pain threshold (PT) was evaluated using an analog algometer (Figure 1). The pain sensitivity was measured on the forearm using two mechanical pain stressors, which indicate which of an ascending sensory stimulus is first perceived as painful. This device is a force gauge that is used to apply an increasing amount of force to the skin through a 1 cm2 surface area until the pain threshold is achieved. This algometer stimulates pain, described as dull pressure at the pain threshold; the reliability and validity of this device have been reported. The pain sensitivity of all measurement patients was taken on the day before the surgery by the same author, and these values were blinded from another author who recorded the repetitive postoperative VAS and knee scores.

Operation Procedure: All patients were operated on in a single-center and experiences in arthroplasty practice. All the patients were operated on standard spinal anesthesia. All patients underwent cruciate-retaining Genesis II knee arthroplasty (Smith and Nephew, Memphis, TN, USA) with a midline incision and medial parapatellar approach with a fixed bearing design. Patella resurfacing was not performed, while patellar denervation was performed in all patients. Bone-cement (40 g) was used with a fourth-generation cementing device.

A pneumatic tourniquet was used before surgery at the proximal thigh and inflated before the skin incision until skin closure in group 1 and no used in group 2. The tourniquet was inflated to either 275 or 325 mmHg, depending on the patient's systolic blood pressure. Peri-operative tranexamic (TXA) acid was administrated intravenously with 20 mg/kg 30 min before surgery. Periarticular injection was not used for pain control in either group. An adductor canal block or epidural analgesia was not applied. Intra-articular drainage was used in every patient, which was removed after 24 h postoperatively.

Postoperative Management and Analgesic Procedure: On the day of surgery, intravenous paracetamol 1 g was given at 8-h intervals, and intramuscular diclofenac sodium 75 mg and intravenous tramadol 100 mg in 100 mL normal saline were given at 12-h intervals. This analgesic procedure was continued at the time of discharge, and all patients were discharged on the third day of surgery. Physical therapy was started on postoperative day 1 in all patients. The functional assessments and range-of-motion were measured during routine physical therapy sessions.

Postoperative Assessment of Pain and Function: VAS score assessment was done at 24 h (rest), 36 h (post-physical therapy), and 48 h (rest) postoperatively. The Knee Society Clinical Scoring System (KSS) was also used for evaluation of functional outcomes, which is a condition-specific validated questionnaire widely used to evaluate the functional capabilities of the knee joint before and after total knee arthroplasty. The KSS was done in the first year postoperatively. The KSS consists of two parts. One part is the knee score (KSS1), which includes pain (maximum 50 points), stability, total range of flexion, and other items (varus, valgus, extension delay, and flexion contracture). The other part (KSS2) is the function score, which has two components, walking capacity and stair-climbing ability and deductions done if the patient using any assistive devices.

ELIGIBILITY:
Inclusion Criteria:

* primary knee osteoarthritis
* older than 18 years
* primary knee arthroplasty

Exclusion Criteria:

* Patients with a neurological disorder,
* diagnosed with fibromyalgia,
* history of knee operation,
* valgus knee,
* greater than 30° flexion contracture
* undergone bilateral knee arthroplasty or revision knee arthroplasty,
* chronic analgesic users, a
* patient with psychiatric disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-06-15 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale Outcome-1 | 24 hour
  Both groups were also evaluated with Visual Analog Scale for assess the pain status postoperatively.
Visual Analog Scale Outcome-2 | 36 hour
  Both groups were also evaluated with Visual Analog Scale for assess the pain status postoperatively.
Visual Analog Scale Outcome-3 | 48 hour
  Both groups were also evaluated with Visual Analog Scale for assess the pain status postoperatively.
Knee Society Score | First year
  The Knee society score (KSS) consists of two parts. One part is the knee score (KSS1), which includes pain (maximum 50 points), stability, total range of flexion, and other items (varus, valgus, extension delay, and flexion contracture). The other part (KSS2) is the function score, which has two components, walking capacity and stair-climbing ability and deductions done if the patient using any assistive devices.

CONTACTS AND LOCATIONS:
Locations (1):
- Umraniye Training and Research Hospital, Istanbul, Umraniye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No